CLINICAL TRIAL: NCT05584865
Title: The Clinical Outcome of Full Digital Fabricated Ocular Prosthesis Versus Conventional Fabricated Technique (a Randomized Controlled Clinical Trial)
Brief Title: Full Digital Fabricated Ocular Prosthesis Versus Conventional Fabricated Technique
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hams Hamed Abdelrahman (Other)
Responsible Party: Sponsor-Investigator, Hams Hamed Abdelrahman, Assistant lecturer of DPH and Clinical statistician, Alexandria University
Organization: Alexandria University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: digital prosthesis_2022
Record Dates: First submitted 2022-10-14; First posted 2022-10-18 (Actual); Last update posted 2022-10-18 (Actual); Status verified 2022-10

CONDITIONS: Occluar Prosthesis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group I (Experimental)
  Interventions: Other: Digital occluar prosthesis
- Group II (Active Comparator)
  Interventions: Other: Conventional occluar prosthesis

INTERVENTIONS:
Other: Digital occluar prosthesis — Each patient will receive the full digital fabricated ocular prosthesis. DICOM data from the Computerized Tomography (CT) will be imported into Materializes Interactive Medical Image Control System (MIMICS) software++++ tool for visualizing and segmenting medical images (such as CT and MRI)
  Arms: Group I
Other: Conventional occluar prosthesis — An accurate impression of the patient's eye socket will be obtained to prepare a suitable wax mod. The wax model will be flasked and processed into heat cured acrylic resin of the same colour of the sclera of the other healthy eye of the patient
  Arms: Group II

SUMMARY:
Different techniques of fabricating conventional custom-made ocular prosthesis were described. Traditional methods of custom fabricated ocular prosthesis had some limitations and take a long time, facial scanning and computed tomography will facilitate the full digital ocular prosthesis fabrication. Full digital ocular prosthesis is an innovated new technique to produce more accurate & more esthetic ocular prosthesis with less time consumed, however very few articles are available comparing between the full digital technique & the conventional one in manufacturing ocular prosthesis.

ELIGIBILITY:
Inclusion Criteria:

* Have enough ocular bed to accommodate the ocular prosthesis.
* At least 3 months after surgery to allow complete healing of the socket.

Exclusion Criteria:

* Patients under steroid therapy or those under radio or chemotherapy.
* Patients having eye lid deformity.
* History of psychological disorder.
* systemic disease.
* eye infection.

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2022-11-01 (Estimated); Primary Completion 2023-05-01 (Estimated); Study Completion 2023-05-01 (Estimated)

PRIMARY OUTCOMES:
Motility of ocular prosthesis | Time of insertion
  Using Matlab R2016b software+. For each patient, photos of different eye positions will be taken, namely, the frontal, upper, lower, left, and right viewing positions.
Change in patient satisfaction | Time of insertion and 3 months
  Patient satisfaction will be evaluated by questionnaire based on the UK National Artificial Eye Questionnaire (NAEQ). The items that will be evaluated in the questionnaire include Time taken to adjust the prosthesis, Prosthesis cleaning frequency, Lubrication frequency, Comfort rating, satisfaction with prosthetic appearance, and satisfaction with prosthetic motility
change in microbial analysis | Time of insertion and 3 months
  Patients will attend 2 visits (0,3 month), in which swab will be collected from the internal surface of the ocular prosthesis as well as from the anophthalmic cavit

CONTACTS AND LOCATIONS:
Locations (1):
- Alexandria Faculty of Dentistry, Alexandria, Egypt

REFERENCES:
- [Derived] Tahmawy YA, Mohamed FS, Elfeki S, Abd-Ellah ME. Microbiological evaluation of conjunctival anopthalmic flora after using digital 3D-printed ocular prosthesis compared to conventional one: a randomized clinical trial. BMC Oral Health. 2023 Dec 18;23(1):1012. doi: 10.1186/s12903-023-03746-w. PMID 38110937